CLINICAL TRIAL: NCT07107061
Title: Pilates and Aerobic Training on Body Composition in Young Adults: a Randomized Controlled Trial
Brief Title: PILATES AND AEROBIC TRAINING ON BODY COMPOSITION IN YOUNG ADULTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Raphael Goncalves de Oliveira, Professor, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GPASD_001_2025
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Improved Body Composition
MeSH Terms: interventions — Exercise; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researcher responsible for randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates (Experimental): A total of 13 exercises were selected for the Pilates group, including two stretching exercises and 11 strengthening exercises for the main muscle groups. Mat exercises and equipment exercises (Ladder Barrel, Cadillac, Step Chair, Reformer, Springboard, and Small Barrel) will be used. Two protocols will be adopted for progression (protocol 1: weeks 1-6; protocol 2: weeks 7-12). Two sets of 10 repetitions will be performed, with a 30-second rest between sets and exercises. The two-by-two rule will be used to increase the load. In this case, the load will increase when the participant performs ≥ 2 repetitions above their target of 10 repetitions in the last set, in two consecutive training sessions. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Pilates exercises
- Aerobic (Experimental): The aerobic group will perform walking/running exercises on a treadmill using the extensive interval training method. To define the intensity and periodization of the training, the running speed associated with V̇O2max (vV̇O2max), second ventilatory threshold (vLV2), and average speed between vV̇O2max and vLV2 (v50%Δ) will be used as reference. These parameters will be obtained from a maximal exercise test on a treadmill, performed before the start of the interventions. Two protocols will be adopted, with adjustments in density (work-to-recovery ratio) every two weeks. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Aerobic exercise
- Pilates plus aerobic (Experimental): They will perform the same exercises as the Pilates group, however, with 1 set of 10 repetitions, with a 30-second rest between sets and exercises, totaling 30 minutes of intervention per session. In the second half of the intervention period, aerobic exercises will be performed, identical to those of the aerobic group, but for 30 minutes. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Pilates exercises plus aerobic exercise
- Control (No Intervention): This group will be instructed to maintain their usual routine.

INTERVENTIONS:
Other: Pilates exercises plus aerobic exercise — Pilates exercises are characterized as muscle strengthening and stretching, while aerobic exercises are characterized as a modality that works cardiorespiratory fitness.
  Other Names: Pilates; aeróbio
  Arms: Pilates plus aerobic
Other: Pilates exercises — Pilates exercises are characterized as muscle strengthening and stretching.
  Other Names: Pilates
  Arms: Pilates
Other: Aerobic exercise — Aerobic exercises are characterized as a modality that works cardiorespiratory fitness.
  Other Names: aerobic
  Arms: Aerobic

SUMMARY:
Pilates exercises have been shown to be effective for a range of outcomes; however, it is unclear whether they can effectively contribute to fat mass reduction, especially when compared with a technique known to be effective for this purpose, such as aerobic training. Furthermore, Pilates' potential for increasing lean mass also requires further investigation. The aim of this study was to assess the effectiveness of Pilates compared with aerobic training, as well as the combination of these activities, on body composition in young adults. Eighty women aged 18 to 40 years were randomized to four groups: Pilates (n = 20), aerobic (n = 20), Pilates plus aerobic (n = 20), and control (n = 20). Body composition was assessed by dual-energy X-ray absorptiometry (DXA), considering: total fat mass (kg), percentage of total fat mass (%), total lean mass (kg), and total lean mass adjusted for height (kg/m²). Additionally, total body mass (kg) and body mass index (BMI) (kg/m2) values were considered. The interventions were carried out for 12 weeks, three times a week, lasting 60 minutes/session. Analyses were performed by intention-to-treat and per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age between 18 and 40 years;
* Not having exercised in the last 6 months;
* Agreeing not to perform any other type of exercise during the study period;
* Being fit to exercise according to the Physical Activity Readiness Questionnaire (PAR-Q) criteria;
* Not having musculoskeletal or neurological disorders that could affect exercise performance;
* Not having known cardiovascular or respiratory diseases;
* Not having cognitive impairment that leads to the inability to follow simple commands;
* Not being a smoker;
* Not being pregnant;
* Not being on any specific diets.

Exclusion Criteria:

* Refusing to sign the informed consent form;
* Unable to complete the pre-intervention assessment procedures.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Percentage of total body fat mass (%) | Baseline and after 12 weeks
  Percentage of total body fat mass assessed by dual-energy X-ray absorptiometry (DXA)
Total lean mass (kg) | Baseline and after 12 weeks
  Absolute total body lean mass assessed by dual-energy X-ray absorptiometry (DXA)
Total fat mass (Kg) | Baseline and after 12 weeks
  Absolute total body fat mass assessed by dual-energy X-ray absorptiometry (DXA)
Total lean mass adjusted for height (kg/m²) | Baseline and after 12 weeks
  Total lean mass adjusted for height assessed by dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Trunk fat mass (kg) | Baseline and after 12 weeks
  Trunk fat mass assessed by dual-energy X-ray densitometry (DXA)
Upper limb fat mass (kg) | Baseline and after 12 weeks
  Upper limb fat mass assessed by dual-energy X-ray densitometry (DXA)
Lower limb fat mass (kg) | Baseline and after 12 weeks
  Lower limb fat mass assessed by dual-energy X-ray densitometry (DXA)
Trunk lean mass (kg) | Baseline and after 12 weeks
  Trunk lean mass assessed by dual-energy X-ray absorptiometry (DXA)
Upper limb lean mass (kg) | Baseline and after 12 weeks
  Upper limb lean mass assessed by dual-energy X-ray absorptiometry (DXA)
Lower limb lean mass (kg) | Baseline and after 12 weeks
  Lower limb lean mass assessed by dual-energy X-ray absorptiometry (DXA)
Total body mass (kg) | Baseline and after 12 weeks
  Total body mass assessed by precision scale
Body mass index (kg/m²) | Baseline and after 12 weeks
  Body mass index calculated by the ratio of total body mass (measured by a precision scale) to height (measured by a stadiometer) squared

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be provided as supplementary material when the study results are published.
Supporting Information: SAP
Time Frame: Between 09/01/2025 until the date of publication of the study.
Access Criteria: The information will be freely accessible.